CLINICAL TRIAL: NCT07112729
Title: A Randomized Controlled Trial Evaluating the Effectiveness of SMS Invitations to Increase Colorectal Cancer FIT Screening Rates Among 45-49-Year-Old Residents
Brief Title: Effectiveness of SMS Invitation on Colorectal Cancer Screening on 45-49-Year-Olds
Acronym: SMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Yueh-Hsia Chiu, Director of Department of Health Care Management, College of Management, Chang Gung University, Principal Investigator, Epidemiology Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202500921B0
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: No Condition
Keywords: Colorectal Cancer Screening; SMS (Short Message Service); Mobile Health (mHealth); Randomized Controlled Trial; Fecal Occult Blood Test (FIT)

STUDY DESIGN:
Intervention Model Description: * Intervention Group (Active SMS Invitation): Participants in this group will receive a text message inviting them to participate in the free FOBT program. The SMS message will include a brief explanation of the program, instructions on how to obtain a screening kit, and a contact number for inquiries. A reminder SMS message will be sent one week after the initial message.
  * Control Group (Standard Notification): Participants in this group will receive the standard notification procedures typically used to inform residents about the FOBT program. After one month of the first SMS sent to the Intervention Group, the Control group will receive the same SMS message as the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active SMS Invitation) (Experimental): Participants in this group will receive a text message inviting them to participate in the free FOBT program. The SMS message will include a brief explanation of the program, instructions on how to obtain a screening kit, and a contact number for inquiries. A reminder SMS message will be sent one week after the initial message.
  Interventions: Other: Active SMS Invitation
- Control Group (No Intervention): Participants in this group will receive the standard notification procedures typically used to inform residents about the FOBT program. After one month of the first SMS sent to the Intervention Group, the Control group will receive the same SMS message as the intervention group.

INTERVENTIONS:
Other: Active SMS Invitation — Participants in this group will receive a text message inviting them to participate in the free FOBT program. The SMS message will include a brief explanation of the program, instructions on how to obtain a screening kit, and a contact number for inquiries. A reminder SMS message will be sent one week after the initial message.
  Arms: Intervention Group (Active SMS Invitation)

SUMMARY:
The goal of this study is to learn if sending text message invitations increases participation in colorectal cancer screening among 45-49 year olds in Yingge District, New Taipei City. It will also assess the effectiveness of this method. The main questions it aims to answer are:

•Does sending text message invitations increase the number of residents who complete fecal occult blood test (FOBT)? This study will compare a group receiving text message invitations to a control group receiving standard notifications to see if text messages are an effective way to increase screening rates.

Participants will:

* Be randomly assigned to either receive text message invitations or standard notifications.
* The intervention group will receive an initial text and a reminder text one week later.
* The control group will receive standard notifications, and after one month will receive the same text message.
* The study will track who obtains a FOBT kit and who completes the test within a three-month period.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to evaluate the effectiveness of active SMS (Short Message Service) invitations for increasing participation in colorectal cancer screening among residents aged 45-49 in Yingge District, New Taipei City.

Background: Colorectal cancer is a significant public health concern, and early detection through screening is crucial for improving outcomes. This study aims to explore a simple and cost-effective method to increase screening rates in a specific population group (45-49 years old) where screening just initiated.

Objectives: The primary objective is to assess whether sending active SMS invitations increases the rate of fecal occult blood test (FOBT) completion among the target population.

Study Design: The study employs parallel randomized controlled trial design.

Eligible participants will be randomly assigned to one of two groups:

* Intervention Group (Active SMS Invitation): Participants in this group will receive a text message inviting them to participate in the free FOBT program. The SMS message will include a brief explanation of the program, instructions on how to obtain a screening kit, and a contact number for inquiries. A reminder SMS message will be sent one week after the initial message.
* Control Group (Standard Notification): Participants in this group will receive the standard notification procedures typically used to inform residents about the FOBT program. After one month of the first SMS sent to the Intervention Group, the Control group will receive the same SMS message as the intervention group.

Intervention:

The contents of SMS is "大腸癌年輕化！國家新政策，符合45-49歲，歡迎參加公費糞便潛血篩檢，顧健康自己來。即日起至8/31止，週一~五8:30-11:30至本所可領採檢管或諮詢電話:098176819鶯歌衛生所關心您。 In English: "Colorectal cancer is affecting younger people! Under a new national policy, those aged 45-49 are welcome to participate in government-funded fecal occult blood screening to take charge of their own health. From now until August 31st, Monday to Friday between 8:30 AM and 11:30 AM, you can visit our office to pick up a collection tube. For inquiries, please call: 0981-768-19 - Yingge Health Center cares about you."

Recruitment: Participants will be identified through the health department's information system, which contains records of residents eligible for the national colorectal cancer screening program and their mobile phone numbers. There is no separate recruitment or enrollment procedure.

•Sample Size: A total of 6,708 eligible residents will be randomly assigned to the intervention and control groups. The sample size is calculated based on previous research, which indicates that approximately 13.1% of individuals in this age group participate in FOBT screening without active intervention. The study aims to increase participation by 5%, reaching an 18% participation rate with SMS invitations.

Timeline: The study will be conducted over from August 5, 2025 to Sep 18, 2025.

Data Collection and Management:

* The health department will provide a de-identified list of eligible residents, including a random code, gender, age, and mobile phone number. This information will be used for random assignment and statistical analysis.
* Random assignment will be performed using computer-generated random numbers.
* The SMS messages will be sent by a contracted SMS provider. The health department will provide the SMS provider with a secure file containing the random code and mobile phone number for each participant.
* The SMS provider will provide data on message delivery status. The health department staff will record whether participants obtain the screening kit and whether they completed fecal occult blood test. This information will be provided to the principal investigator (PI) for analysis.

Outcome Measures:

•Primary Endpoint: Numbers of completed fecal occult blood test. Data Analysis: The primary analysis will be conducted using an intention-to-treat (ITT) approach, where all participants will be included in the analysis based on their assigned group, regardless of whether they received the intervention or completed the screening.

Ethical Considerations: The study has been designed to protect the privacy and confidentiality of participants. Data will be de-identified and stored securely. All personal data will be protected through anonymized coding and data encryption. SMS dissemination will be handled by a third-party vendor under confidentiality agreements, and no personally identifiable information will be shared beyond phone number use for message delivery. The project is funded through existing administrative cancer screening budgets, without external sponsorship. The study will comply with all relevant ethical guidelines and regulations.

ELIGIBILITY:
Inclusion Criteria:

* Residents aged 45-49 in Yingge District, New Taipei Cit
* Must have registered mobile numbers

Exclusion Criteria:

* Not resident in Yingge District
* Age not in 45-49
* Without registered mobile phone numbers

Ages: 45 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6708 (Actual)
Dates: Start 2025-08-07 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | From first SMS to 31 days
  Number of participants who Completed the fecal occult blood test. The date after SMS invitation of FIT completed was collected for evaluation with observed period (31 days).

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Yueh-Hsia CHIU, PhD, Principal Investigator — Department of Health Care Management, Chang Gung University
Locations (1):
- Yingge District Public Health Center, New Taipei City, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Based on research collaboration, de-identified participant-level results can be required from Principal Investigator.
Supporting Information: SAP
Time Frame: 2027/1/1-2029/12/31
Access Criteria: Based on research collaboration and request by email.